CLINICAL TRIAL: NCT00587184
Title: The Use of Confocal Microscopy in Barrett's Esophagus
Brief Title: Confocal Microscopy in Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenneth K. Wang, VanCleve Professor of Gastroenterology Research, Mayo Clinic
Other Study IDs: 06-004664
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2013-11

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Confocal Microscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients who were seen clinically indicated endoscopic surveillance and biopsies of BE and confocal microscopy was performed.

SUMMARY:
This data review will be done to evaluate the use of confocal microscopy imaging in patients who were seen for clinically indicated endoscopic surveillance and biopsies of Barretts Esophagus

DETAILED DESCRIPTION:
This retrospective chart review will be done to evaluate the use of confocal microscopy imaging in patients who were seen at Mayo Clinic for clinically indicated endoscopic surveillance and biopsies of BE.

Endoscopy reports and pathology results will be reviewed from 100 patients who have undergone endoscopy. These results will be correlated with images obtained with confocal microscopy at the time of the endoscopy. There will be no patient contact.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone confocal microscopy at the time of surveillance endoscopy for Barrett's Esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had confocal microscopy imaging in patients at the time of or clinically indicated endoscopic surveillance and biopsies of BE.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2006-07; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States